CLINICAL TRIAL: NCT00157521
Title: A Double-Blind, Randomized, Pilot Study to Explore Whether Enhancing L-Arginine Bioavailability by Oral Supplementation Increases NO Production and Prevents Peroxynitrite Generation in the Pre-Eclamptic Placenta
Brief Title: L-Arginine in Pre-Eclampsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: L-ARG
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Arginine

INTERVENTIONS:
Drug: L-arginine

SUMMARY:
Pre-eclampsia is a disorder unique to pregnancy affecting both the mother and the fetus. Hypertension, proteinuria and edema are the most common and well-known maternal clinical symptoms. The incidence is approximately 6-8%. Pre-eclampsia is one of the leading causes of maternal and fetal mortality and morbidity associated with pregnancy throughout the world. The pathophysiology is unknown. At present, the most effective treatment is immediate delivery.

The researchers' studies contributed to the demonstration that the vasodilator nitric oxide (NO) is important for correct placentation and that less nitric oxide (NO)- dependent vasodilation and an excess formation of reactive oxygen species explain poor placenta perfusion in pre-eclampsia. This reduced NO activity and increased oxidative stress in pre-eclamptic placenta is related to low bioavailability of L-arginine, the NO precursor.

In this pilot study the researchers want to evaluate whether the administration of L-arginine to women with a clinical diagnosis of preeclampsia might restore physiological NO production in the placenta and ameliorate the pregnancy outcome.

DETAILED DESCRIPTION:
INTRODUCTION

In the past few years evidence has accumulated strongly suggesting that nitric oxide (NO), a potent endothelial-derived vasodilator, might be implicated in gestational vasodilatation. NO is synthesized from the aminoacid L-arginine by a family of enzymes, the NO synthases (NOS). The endothelial isoform of nitric oxide synthase (ecNOS) has been found in the human placenta and immunohistochemically localized to the endothelium of the umbilical cord, chorionic plate and stem villous vessels. Locally formed ecNOS-dependent NO may serve to maintain low vascular resistance besides attenuating the action of vasoconstrictors. With its unique angiogenic/vasculogenic properties, NO can be instrumental for promoting cytotrophoblast endovascular invasion of uterine spiral arteries, an essential feature of normal placentation. Inadequate production of the vasodilator nitric oxide (NO) in the placenta has been recently suggested to explain the high resistance state and the ineffective placentation of pre-eclampsia, however the results to date are conflicting. We recently found that placental endothelial NO synthase (ecNOS) expression and activity were comparable in normal pregnancy and in pre-eclampsia, but in pre-eclamptic placenta NO is degraded to peroxynitrite, that is good candidate for mediating the oxidative damage of pre-eclampsia. Concentration of the NO precursor L-arginine was lower in pre-eclampsia, suggesting a defect in L-arginine bioavailability in the placentas. These results provide a biochemical explanation for the defective NO synthesis in pre-eclamptic placenta since NO production by endothelial NO synthase (ecNOS) is strongly dependent on the availability of the substrate L-arginine so that low L-arginine availability induces NOS to synthesize peroxynitrite at the expense of NO.

These results suggest that, in the normal placenta, adequate concentration of L-arginine selectively orients ecNOS toward NO, which is vital for a normal placentation.In the pre-eclamptic placenta, instead, a lower than normal L-arginine concentration re-directs ecNOS toward peroxynitrite which is generated in exuberant amounts at the expense of NO. This favors microvascular damage and impairs cytotrophoblast invasion.

Thus, whether increasing L-arginine bioavailability might restore physiological NO production in pre-eclamptic placenta is worth investigating in a pilot study that might represent the basis of a large, multicenter trial aimed to explore the impact of the above treatment on pregnancy outcome.

AIMS

Primary

* To compare L-arginine and NO metabolite (NO2-/NO3-) concentrations in systemic and umbilical cord blood, and placental ecNOS, nitrotyrosine and HNE-lysine staining and levels of conjugated dienes in ten pre-eclamptic women given L-Arginine supplementation and in ten pre-eclamptic women given placebo.
* To compare L-arginine transport activity in normal and pre-eclamptic placenta syncytiotrophoblasts in vitro. To compare the mRNA expression of cationic aminoacid systems (Y+ LAT, CAT-2 and CAT-4) in normal and pre-eclamptic placenta.

Secondary

* To compare in pre-eclamptic women given L-Arginine supplementation and in pre-eclamptic women given placebo the following:
* Time from pre-eclampsia onset to delivery
* Arterial blood pressure, albuminuria, proteinuria, complete blood cell count including platelet count, serum creatinine, uric acid, triglycerides, cholesterol, C3, GOT, GPT, GammaGT, HDL, LDL and LDH concentration at the time of delivery
* Structural changes of the placenta
* Newborn weight, height, and Apgar score
* Gestational age at delivery

DESIGN

Ten women with clinical diagnosis of pre-eclampsia given oral L-arginine supplementation from the time of diagnosis (cases) and ten women with clinical diagnosis of pre-eclampsia on placebo (controls) matched with cases for age, parity, time of onset of pre-eclampsia and concomitant risk factors (chronic hypertension, diabetes, renal disease, multiple pregnancy) will be selected for study participation. Cases and controls will also receive conventional therapy (antihypertensive drugs: nifedipine, alpha-methyldopa; magnesium for prophylaxis of eclampsia; betamethasone for fetus maturation) for pre-eclampsia and will be homogenous for treatment. Ten normotensive pregnant women (normotensive pregnancy) matched for gestational age and for type of delivery (cesarean or vaginal) will be also studied. All subjects will provide a written informed consent according to the declaration of Helsinki. Patients will enter the study as soon as diagnosis of pre-eclampsia will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-eclamptic women

   * Pregnancy - induced hypertension (diastolic blood pressure [DBP] ≥ 90 mm Hg) and
   * Proteinuria ≥ 300 mg/24 h or albuminuria ≥ 250 µg/min and/or
   * Early signs of intrauterine growth restriction (IUGR) more than 2 standard deviations below the mean for gestational age in patients with a previous ultrasound test before 20th week of gestation
2. Normotensive pregnant women

   * Diastolic blood pressure < 90 mm Hg
   * No history of hypertension
   * No significant proteinuria
   * No signs of infection
   * No signs of IUGR
   * Matched for gestational age with pre-eclamptic women

Exclusion Criteria:

* History of hypersensitivity to l-arginine
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of trial
* Evidence of uncooperative attitude
* Any evidence that allows predicting that the patient will not be able to complete the trial follow-up

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2002-09; Study Completion 2006-05

PRIMARY OUTCOMES:
NO production, at delivery

SECONDARY OUTCOMES:
Pregnancy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Principal Investigator — Mario Negri Institute
Locations (2):
- Italy (2):
  - Hospital "Ospedali Riuniti", Unit of Obstetrics and Ginecology, Bergamo, Bergamo
  - Obstetrics and Ginecology Division, Brescia